CLINICAL TRIAL: NCT06013150
Title: A Phase 1, 2-Part Study in Healthy Male and Female Participants; Part 1 - A Randomised, Double-Blind, Placebo-Controlled, Single Ascending Dose-Escalation Study of Inhaled DMC-IH1; Part 2 - An Open-Label, 3-Arm Study Assessing the Carryover Effects of Inhaled (DMC-IH1) and Intramuscular (EpiPen®) Epinephrine
Brief Title: Study of Inhaled DMC-IH1 and Intramuscular (EpiPen®) Epinephrine in Healthy Male and Female Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: De Motu Cordis (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DMC-CL-002
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Anaphylactic Reaction
MeSH Terms: conditions — Anaphylaxis | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine (Experimental): Dosage Level:
  Part 1 of the study: Participants across cohort 1 to 3 will receive a single dose of either 1mg or 1.3mg or 1.5mg respectively of epinephrine or placebo via DMC-IHI device.
  Dosage form: Single-use capsule based dry powder inhaler
  Route of administration: Inhalation
  Interventions: Drug: Epinephrine; Drug: Placebo
- Placebo (Placebo Comparator): Drug: Placebo
  Participants will receive matching placebo across the study.
  Interventions: Drug: Epinephrine; Drug: Placebo

INTERVENTIONS:
Drug: Epinephrine — Participants in Part 1 of the study will receive single dose either 1mg, 1.3mg or 1.5mg of an inhaled single dose of Epinephrine or placebo delivered via DMC-IHI device.
Drug: Placebo — Participant in Part 1 of the study will receive matching doses of placebo

SUMMARY:
This is a phase 1, randomised, double blind placebo controlled 2-part study to assess the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of inhaled DMC-IH1 (epinephrine) and relative bioavailability and carryover effects of Inhaled (DMC-IH1) and Intramuscular(IM) (EpiPen®) Epinephrine in healthy male and female participants.

DETAILED DESCRIPTION:
DMC-IH1 (Investigational product) inhaler is a proprietary single-use capsule based dry powder inhaler designed for oral pulmonary drug delivery in emergency scenarios.

Part 1 will enrol 24 participants into 3 cohorts receiving a single ascending dose.

Study will comprise 3 periods: Screening, Treatment Period and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing to sign an ICF on a voluntary basis and to voluntarily participate in the study, after being able to read the ICF and understand the information contained within, prior to any Screening procedure being undertaken.
2. Male or female and ≥18 to ≤45 years of age at time of signing the ICF.
3. Has a BMI of ≥18.00 to ≤30.00 kg/m2, with a minimum body weight of 45.0 kg and a maximum body weight of 120 kg.
4. Is in good health based on the results of medical and surgical history, physical examination, vital sign measurements, and clinical laboratory evaluations, as assessed by the Investigator (or designee).
5. Has a resting heart rate of ≥45 and ≤90 beats per minute; systolic blood pressure of ≥90 but ≤130 mmHg and diastolic blood pressure of ≥50 but ≤90 mmHg at Screening (Visit 1) and prior to randomisation on Day -1 (Visit 2).
6. Has normal lung function assessed using spirometry and defined by forced vital capacity (FVC) ≥ lower limit of normal (LLN), forced expiratory volume in 1 second/FVC ≥LLN, and peak inspiratory flow rate ≥ LLN at Screening (Visit 1).
7. Has no history of anaphylaxis or severe allergy requiring the use of epinephrine.
8. Is a non-smoker/non-vaping; or social smoker who currently only uses ≤5 cigarettes per month and has used nicotine on ≤5 occasions within 30 days prior to Screening, a negative cotinine test at Visit 2/Day -1, and ability and willingness to refrain from smoking 7 days prior to the first epinephrine dose through the EOS [Part 1: Visit 3].
9. Has adequate venous access.
10. Is able to demonstrate correct use of the device using a practice device and follow directions for use.
11. Able to follow contraceptive measures as per Protocol.
12. Ability and willingness to refrain from undertaking any strenuous exercise (including weightlifting) 48 hours prior to each clinic visit.
13. Ability and willingness to refrain from alcohol and/or drug use from Screening (or at least 1 week prior to dosing) (testing at Day -1 to ensure compliance) until EOS (Part 1: until Visit 3/EOS).

Exclusion Criteria:

1. Participant who is pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time from screening to the end of study visit (Part 1: through Visit 3/EOS).
2. Participant has a history of significant hypersensitivity or intolerance to lactose and/or epinephrine.
3. Participant has a history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular (including severe pulmonary haemorrhage), gastrointestinal, neurological (including history of migraine requiring specific treatment), respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee) except for fully resolved childhood asthma.
4. Participant has a positive urine drug screen at Screening and at Baseline (Visit 2/Day -1).
5. Participant has a positive urine cotinine test at Baseline (Visit 2/Day -1).
6. Participant took part in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to Baseline (Visit 2/Day -1).
7. Participant used or intends to use any prescription or non-prescription medications/products within 14 days prior to randomization (Day -1) through EOS (Part 1: Visit 3/EOS), with the exception of paracetamol/acetaminophen at the discretion of the Investigator, and contraceptives.
8. Participant has a history of alcoholism or substance or drug abuse-related disorders deemed significant by the Investigator (or designee) (ie, >14 drinks/week for women or >21 drinks/week for men [1 drink=150 mL of wine or 360 mL of beer or 45 mL of hard liquor]) within the last 3 months prior to Screening (Visit 1) and randomization (Day -1/Visit 2).
9. Participant has a positive alcohol breath test at Screening and prior to randomization (Day -1/Visit 2).
10. Female participant has a positive serum pregnancy test at Screening and a positive urine pregnancy test prior to randomization (Day -1/Visit 2).
11. Participant has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C virus antibody (anti-HCV) with HCV RNA detected at Screening and hepatitis B core antibody at Screening.
12. Participant has presence of any physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
13. Participant has received any of the following vaccinations:

    1. Live vaccine(s) within 1 month prior to Screening or plans to receive such vaccines during the study.
    2. Killed vaccine 1 week prior to randomization (Day -1/Visit 2).
    3. COVID-19 vaccine Day -7 through Visit 3 for Part 1.
14. Participant had surgery of the nose/paranasal sinuses/mouth/throat within 8 weeks or thoracic surgery within 24 weeks prior to Screening or randomization (Day -1/Visit 2).
15. Participant has any history of clinically relevant respiratory (especially with reduction of respiratory capacity) or history of clinically significant cardiovascular abnormality (eg, including hypertension, ischemic heart disease, previous myocardial infarct, heart failure or conduction abnormalities (SVT, AF, interventricular conduction blocks, etc.) or any other abnormality that in the opinion of the Investigator may pose a safety risk to a participant), or any other abnormality that in the opinion of the Investigator may pose a safety risk to a participant in this study may confound the clinical performance or safety assessment, or may interfere with study participation.
16. Participant has any of the following ECG criteria:

    1. PR interval >220 ms or <120 ms
    2. QRS interval >120 ms
    3. QTcF interval >450 ms (males) or >470 ms (females)
    4. A marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval >450 ms)
    5. ST segment elevation or depression considered to be clinically significant by the PI or designee
    6. T-wave or U-wave abnormalities considered to be clinically significant by the PI or designee -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Upto 7 days for Part 1
Number of participants with clinical laboratory abnormalities | Upto 7 days for Part 1
Number of participants with changes in the 12-lead electrocardiogram (ECG) | Upto 7 days for Part 1
PK Parameters: Assess timepoints of carryover effect of repeated dose of inhaled epinephrine | Part 1: Pre-dose and multiple timepoints post dose on Day 1.

SECONDARY OUTCOMES:
PK Parameters: Time for maximum concentration (Tmax) | Part 1: Pre-dose multiple timepoints post-dose on Day 1.
PK Parameters: Maximum concentration (Cmax) | Part 1: Pre-dose multiple timepoints post-dose on Day 1.
PK Parameters: Area under Curve (AUC) | Part 1: Pre-dose multiple timepoints post-dose on Day 1.
PD parameters: Maximum effect on heart rate and blood pressure (Emax) | Part 1: 240 minutes postdose.
PD parameters: Time to maximum effect (TEmax) | Part 1: 240 minutes postdose.

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Neil, Study Director — peter.oneill@demotucordis.co
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No